CLINICAL TRIAL: NCT01806727
Title: Lifestyle Intervention for Treatment of Diabetes
Acronym: LIFTDiabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00022613; 1P60MD006917-01 (NIH)
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes; Overweight; Obesity
Keywords: Diabetes; Diabetes Self Management; LIFT Diabetes; Weight Loss; Diet; Physical Activity; Overweight; Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Diabetes Mellitus; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Self Management (DSM) (Active Comparator): Diabetes Self Management education, delivered in the clinics, using group-based visits and targeting improved control of hemoglobin A1c and related risk factors.
  Interventions: Behavioral: Community Lifestyle Weight Loss (LWL)
- Community Lifestyle Weight Loss (LWL) (Experimental): Participants with type 2 diabetes will be enrolled in a 12 month lifestyle intervention designed to achieve a mean >7% weight loss induced through caloric restriction and increased physical activity. The intervention will be delivered via supervised Community Health Workers (CHWs). Most meetings will be at a community location.
  Interventions: Behavioral: Diabetes Self Management (DSM)

INTERVENTIONS:
Behavioral: Community Lifestyle Weight Loss (LWL) — Changing dietary and physical activity behavior to promote weight loss
  Arms: Diabetes Self Management (DSM)
Behavioral: Diabetes Self Management (DSM) — Changing diet, physical activity, self monitoring, and medication related behaviors to improve diabetes control
  Arms: Community Lifestyle Weight Loss (LWL)

SUMMARY:
This study is evaluating two approaches to improving the control blood sugar, and other risk factors for heart disease in overweight and obese adults with type 2 diabetes. The first approach has participants focus on weight loss via reducing food intake and increasing physical activity, while attending weekly group sessions led by trained community health workers for 12 months. The second approach has participants receive education on diabetes self management, which focuses primarily on glucose control, while attending monthly group sessions led by a study staff member for 12 months. We are recruiting persons with type 2 diabetes who live in the Winston-Salem/Forsyth County area of North Carolina who are willing to attend sessions at the Downtown Health Plaza of Wake Forest Baptist Health. We will measure risk factors for heart disease (glucose control, blood pressure, blood cholesterol) and calculate the predicted risk of heart disease, and see which intervention lowers risk to a greater extent at 12 months, as well as 24 months.

DETAILED DESCRIPTION:
The Look AHEAD trial has demonstrated improved risk factor control among overweight or obese diabetes patients who received an intensive lifestyle intervention at both one and four years after enrollment. Translating such findings into accessible and effective weight loss programs is a major public health challenge. We are conducting "Lifestyle Interventions for Treatment of Diabetes" (LIFT Diabetes). The overall goal is to investigate two approaches to improving risk factor control; one which is modeled after Look AHEAD and is designed to achieve 7% weight loss and increase physical activity to > 175 minutes per week among minority and lower income diabetes patients via a 12-month, group based lifestyle intervention, using community health workers supervised by an interventionist. Participants will have up to 4 group visits/month and up to 12 individual contacts/year. The other approach will promote Diabetes Self Management (DSM) by educating participants regarding health behaviors which lead to improved diabetes control; this arm is also 12 months, and is delivered in the clinic by intervention staff via monthly group visits and up to 12 individual contacts/year. We will randomize 260 overweight or obese adults with diabetes to either intervention, and determine the impact on outcomes (UKPDS-estimated CVD risk, risk factor control), weight, cost, resource utilization, and safety at 12 months, and after transitioning back to usual care, at 24 months. The hypotheses are that the community based intervention results in 10% relative reduction in CVD risk compared to clinic-based intervention; the interventions are equivalent with respect to adherence and participant satisfaction; and the community based intervention is associated with lower cost than the clinic based intervention. Translating evidence based, lifestyle strategies, and targeting minority and underserved patients, will yield, if successful, models for addressing diabetes-related health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 21 years of age and older residing in the Forsyth County, North Carolina region.
* Disease: Type 2 diabetes mellitus.
* Overweight or obese: defined as body mass index (BMI) greater than 25 kg/m2 (>27 if on insulin).
* If not on diabetes medication, persons with hemoglobin A1c greater than or equal to 6.5% and less than 11.0%
* If on diabetes medication, hemoglobin A1c greater than or equal to 5.0% and less than 11.0%
* Blood pressure: BP ≤ 160/100 mmHg.
* A usual source of medical care: The intervention may induce hypoglycemia and have other risks, and weight loss and increased physical activity may modify the need for drugs used to treat diabetes, high blood pressure, and lipids. Patients must have a source for ongoing care. Usual source of care will be documented via a "medical clearance" form with physician signature verifying that MD is aware their patient is participating in this trial.
* Able to exercise: Increasing moderate intensity physical activity is an integral part of this intervention. Must be able to walk 1/4 mile without assistance.
* Able to communicate in English
* Other: Willing to give consent to participate in this research program, including random allocation to either study arm.

Exclusion Criteria:

* Poorly controlled diabetes: defined by hemoglobin A1c>11%
* Cardiovascular disease: Clinical history of cardiovascular disease, or newly diagnosed at screening. This includes myocardial infarction, heart failure, ischemic heart disease, stroke and other vascular disease. Persons suspected of having angina (chest pain) or other potentially ischemic symptoms will be required to be evaluated by their health care provider.
* Weight Loss: Currently involved in a supervised medical or surgical weight loss program or with a history of prior weight loss surgery.
* Age: We will exclude children (<21 years)
* Pregnancy: Diabetes during pregnancy has specific management criteria, and the role of weight loss via caloric restriction and increased physical activity is of uncertain efficacy and safety. Among women of child-bearing potential, planning to become pregnant within 12 months will be an exclusion criteria. Women who have recently given birth and are breast feeding are also excluded
* Serious Illness with anticipated decreased life expectancy during the 2 year (24 month) time frame of the intervention, such as cancer diagnosis or treatment within the past 5 years (with the exception of non-melanoma skin cancer).
* Inability to exercise: Patients who are wheel chair bound, have had an amputation, are undergoing treatment for lower extremity infections, or who self report being unable to ambulate 400 meters (1/4 mile) without assistance.
* Participation in another clinical trial involving intervention(s) which affect any component of cardiovascular risk. Potential participants who are enrolled in purely observational studies remain eligible.
* Renal disease: Persons with stage 3 chronic renal disease (estimated glomerular filtration rate <60ml/min by the chronic kidney disease formula used by Wake Forest Baptist) will be excluded.
* Other: Conditions/criteria likely to interfere with participation and acceptance of randomized assignment, including the following: inability/unwillingness to give informed consent, major psychiatric or cognitive problems (schizophrenia, dementia), self-reported active illegal substance or alcohol abuse, and clinical judgment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Predicted Cardiovascular Risk | 12 months
  Cardiovascular risk will be estimated by the United Kingdom Prospective Diabetes Study (UKPDS) risk score, which is based on age, gender, diabetes duration, hemoglobin A1c, blood pressure, lipids, and smoking status. The study will compare the mean changes in UKDPS scores between groups at 12 months.

SECONDARY OUTCOMES:
Hemoglobin A1c | 12, 24 months
  Change (from baseline) in HbA1c at 12 and 24 months between groups will be assessed
Blood Pressure | 12, 24 months
  Systolic and Diastolic Blood Pressure change from baseline at 12 and 24 months between groups will be assessed
Lipids | 12, 24 months
  Changes in the lipid profile (Total Cholesterol, HDL-Cholesterol, LDL-Cholesterol, Triglycerides) from baseline to 12 and 24 months between groups will be determined
Weight Change | 12, 24 months
  Change in weight from baseline at 12 and 24 months will be ascertained
Predicted Cardiovascular Risk | 24 months
  24 month change in UKPDS score will be determined and compared across arms.

OTHER OUTCOMES:
Health Costs | 12, 24 months
  Costs and resource utilization will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Alain G Bertoni, MD MPH, Principal Investigator — Wake Forest University Health Sciences; Jeffrey Katula, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Claudel SE, Bertoni AG. Exploring the Use of Personal Technology in Type 2 Diabetes Management Among Ethnic Minority Patients: Cross-Sectional Analysis of Survey Data from the Lifestyle Intervention for the Treatment of Diabetes Study (LIFT Diabetes). JMIR Diabetes. 2018 Feb 22;3(1):e5. doi: 10.2196/diabetes.8934. PMID 30291086
- [Derived] Effoe VS, Katula JA, Kirk JK, Pedley CF, Bollhalter LY, Brown WM, Savoca MR, Jones ST, Baek J, Bertoni AG; LIFT Diabetes Research Team. The use of electronic medical records for recruitment in clinical trials: findings from the Lifestyle Intervention for Treatment of Diabetes trial. Trials. 2016 Oct 13;17(1):496. doi: 10.1186/s13063-016-1631-7. PMID 27733193